CLINICAL TRIAL: NCT05885191
Title: True Ileal Amino Acid Digestibility of Tenebrio Molitor Larvae Determined by Dual Stable Isotope Tracer Method in Young Women
Brief Title: True Ileal Amino Acid Digestibility of Tenebrio Molitor Larvae in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diego Moretti (Other)
Collaborators: Swiss Distance University of Applied Sciences (Other); Swiss Federal Institute of Technology (Other); St. John's Research Institute (Other); Wageningen University and Research (Other)
Responsible Party: Sponsor-Investigator, Diego Moretti, Head of Nutrition Research, Swiss Distance University of Applied Sciences
Organization: Swiss Distance University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TmD01
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Malnutrition; Protein
Keywords: edible insects; Tenebrio molitor; digestibility; protein quality; amino acids
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2H intrinsically-labeled T.molitor (Experimental): 1 portion of bread and vegetable soup prepared with dried 2H intrinsically labeled T.molitor and 13C labeled reference amino acid mixture
  Interventions: Other: 2H intrinsically-labeled T.molitor with 13-C labeled amino acid mixture

INTERVENTIONS:
Other: 2H intrinsically-labeled T.molitor with 13-C labeled amino acid mixture — Test meal with dried 2H intrinsically labeled T.molitor and 13C labeled reference amino acid mixture will be divided into 10 portions, which will be given hourly over the course of 7 hours. The first consumption will be the priming meal, comprised of 3 portions and will additionally contain 13C sodium bicarbonate.

SUMMARY:
Dietary protein intake of adequate quality is essential for human health. Traditional animal source foods play a key role in providing high quality protein but are associated with a high burden on the environment. Therefore, viable alternative protein sources are needed to be able to meet human nutritional needs for the rapidly increasing world population, while keeping food production within the planetary boundaries. T. molitor (Yellow Mealworm larvae) is a sustainably produced and commercially available edible insect, which contains a high quantity of protein with a favorable amino acid profile. Protein quality evaluation considers the amino acid composition as well as the ileal digestibility of the food's individual amino acids, to assess if human dietary requirements for essential amino acids can be met by the protein source. The present study will measure the digestibility of essential amino acids from T. molitor with a minimally invasive dual stable isotope tracer method that follows a plateau-fed test meal protocol. T. molitor will be intrinsically labelled with the stable isotope deuterium (2H), which will be given along with a reference amino acid mixture of known digestibility, labelled with the stable isotope carbon-13 (13C). Based on the results from the present study, protein quality of T. molitor as a protein source for human nutrition can be assessed, allowing a direct comparison of this novel protein source to other protein sources, such as meat and legumes.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18-45 years
* Normal BMI (18.5 - 25 kg/m2)
* Body weight < 60 kg
* Signed informed consent
* Able to communicate and comprehend English
* Are open-minded towards consuming insect-based meals

Exclusion Criteria:

* Anaemic (Hb < 12 g/dL)
* Inflammation (CRP > 5.0 mg/L)
* Pregnancy or intention to become pregnant during the study or within 30 days after the discontinuation of the study intervention
* Lactating up to 6 weeks before the study initiation
* Chronic digestive, renal and/or metabolic diseases
* Antibiotics in the last 4 weeks prior to the study and during the study
* Mineral and vitamin supplementation in the last 2 weeks prior to the study
* Chronic medication intake (except for oral contraceptives)
* Daily exercise routine of high intensity
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Participation in any clinical study within the last 30 days
* Food allergies, especially hypersensitivity to crustacea, dust mites, sea food, gluten, milk, or eggs
* History of serious illness or infection within 3 months of the study
* Cigarette smoking (> 1 cigarette per day)
* Difficulties with blood or breath sampling
* Participants who cannot be expected to comply with study protocol (e.g., not available for the full 8.5 hours of the study day or unable to follow fasting period)
* Inability to understand the information sheet and the informed consent form due to cognitive or language reasons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
True ileal amino acid digestibility | 1st day
  True ileal amino acid digestibility of intrinsically 2H labelled mealworm larvae (Tenebrio molitor) will be determined, relative to a simultaneously administered 13C labelled amino acids mixture, by measuring the plasma appearance of 13C and 2H isotopic enrichments of amino acids at plateau

SECONDARY OUTCOMES:
Hemoglobin (Hb) | -14 days
  Iron status marker
C-Reactive Protein (CRP) | -14 days
  inflammation status
Appearance of 13CO2 enrichment in breath | 1st day
  Rate of amino acid oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, Prof. Dr., Principal Investigator — Swiss Distance University of Applied Sciences
Locations (1):
- ETH Zurich, Laboratory of Human Nutrition, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No